CLINICAL TRIAL: NCT00467064
Title: Arthritis Self-Management Education -- Dose Response
Brief Title: Arthritis Self-Management Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Stanford University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Jean Goeppinger, UNC-Chapel Hill
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 06-0398-1-3; S3521-24/24 (Other Grant/Funding Number: CDC)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Arthritis
Keywords: Disease self-management; Community programs
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthritis self-management workshop (Experimental): Comparison of two-week, lay led, scripted self-management workshop emphasizing action planning, problem-solving, and content specific to arthritis.
  Interventions: Behavioral: Arthritis Quick Start; Other: Delayed treatment intervention
- Delayed treatment control (Other): After 4 month delay, participants in Control Group receive Experimental intervention.
  Interventions: Other: Delayed treatment intervention

INTERVENTIONS:
Behavioral: Arthritis Quick Start — Two week, lay led, workshop focusing on goal setting, problem solving, and content specific to disease management.
  Arms: Arthritis self-management workshop
Other: Delayed treatment intervention — After four months delay, participants in Control Group receive Experimental workshop.

SUMMARY:
We will develop brief versions of the classic 6-week Arthritis Self-Management Program and evaluate their effectiveness.

DETAILED DESCRIPTION:
Many national statements have been made recently about the importance of evidence-based arthritis self-management to improvements in the public's health. The prevalence of arthritis is increasing as the US population ages; the prevalence of arthritis-related disability is higher among Blacks than Whites. Effective arthritis self-management education programs with varying formats have been developed and found effective. Despite this, many Arthritis Foundation chapters and arthritis units of state health departments have found dissemination difficult, and cite the time demands (6 weekly sessions, 2 hours/session) of the classic arthritis self-management education program (ASMP) as a major barrier. Researchers at the University of North Carolina at Chapel Hill and Stanford University will develop and evaluate two "low dose" arthritis self-management programs. The study will be conducted in three phases. Phase One (Development): Researchers will conduct needs assessments with arthritis self-management program disseminators, rheumatologists and other arthritis health professionals, and potential program users to determine preferred content, length, and schedule. Using findings from these assessments, researchers will develop two "low dose" versions of the ASMP. Phase Two (Implementation and Evaluation): Researchers will evaluate the "response" (effectiveness) of both "low dose" interventions in a randomized controlled trial (4 months) and a longitudinal study (one year). We will measure four outcomes: (1) Self-Management Behaviors, (2) Arthritis Self-Efficacy, (3) Health-related Quality of Life (Self-reported Health, Pain, Disability, Fatigue, Activity Limitation, and Health Distress); and (4) Health Care Utilization. A sample of 700 adults with diagnosed arthritis or chronic joint pain, including 200 African Americans, will participate in the study. All data will be gathered via self-administered mailed questionnaires, with telephone follow-up as needed. We will use analysis of co-variance and structural equation modeling to evaluate effectiveness. Researchers will also compare the effectiveness of each new "low dose" program with the effectiveness of existing arthritis self-management education program options. Phase Three (Dissemination): We will consult with arthritis units of state health departments and state chapters of the Arthritis Foundation on program adoption and distribution.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older
* Arthritis diagnosis
* No prior participation in arthritis self-management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2006-10; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | 10-1-05-9-30-09

SECONDARY OUTCOMES:
Self-reported health | 10-1-05-9-30-09

CONTACTS AND LOCATIONS:
Overall Officials: Jean Goeppinger, PhD, BSN, Principal Investigator — University of North Carolina, Chapel Hill; Kate Lorig, DrPH, BSN, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University Patient Education Research Center, Palo Alto, California
  - University of North Carolina Center for Health Promotion & Disease Prevention, Chapel Hill, North Carolina